CLINICAL TRIAL: NCT05963438
Title: Comparison Of En-Masse Retraction With Two-Step Retraction Using Mini-Implant As Anchorage - A Randomized Controlled Trial
Brief Title: Comparison Of En-Masse Retraction With Two-Step Retraction Using Mini-Implant As Anchorage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Anam Sattar, Senior Registrar, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2681
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-02

CONDITIONS: En-masse Retraction to Two- Steps Retraction
Keywords: En-masse retraction, Two step retraction, mini-implant; anchorage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two-step retraction group (control group) (Other): In this group, immediately after placement of mini-implant and extractions of upper first premolars, heavy ligation will be done from mini-implant to maxillary second premolar and first molar. Canine will be retracted by sliding mechanics and the four anterior teeth will be retracted by loop mechanics. Loops will be activated every three weeks by 1 mm.
  Interventions: Procedure: anterior retraction
- En-masse retraction group(experimental group) (Experimental): After placement of mini-implants and extraction of maxillary first premolar, rectangular stainless steel arch wire with anterior 8mm height crimpable hooks distal to the lateral incisors will be inserted and force will be applied using elastic chains attached between the mini-implant and the hooks for conducting en-masse retraction. Elastic chains will replace after every three weeks
  Interventions: Procedure: anterior retraction

INTERVENTIONS:
Procedure: anterior retraction — After placement of mini-implants and extraction of maxillary first premolar, retraction of anterior either simultaneously or separately depending on the allocated group will be done

SUMMARY:
This Randomized Control Trial will be conducted to compare the effects of en-masse retraction to two- steps retraction on sagittal, vertical and dental dimensions using mini-implant as anchorage.

DETAILED DESCRIPTION:
Extractions of teeth are the commonest approach in treating orthodontic problems. There is several extraction protocol commonly employed in the orthodontic correction of class II malocclusion ranging from the extraction of two premolars (20.2%) to four premolars (42.9%).

Retraction of anterior teeth followed by the extraction of premolars requires anchorage to restrict the mesial movement of posterior teeth. Anchorage control is a major factor in achieving successful orthodontic treatment and it can be achieved by variety of appliances, of which titanium screws have been considered as an absolute source of anchorage in orthodontics treatment. The anchorage reinforced from mini-implant is helpful in minimizing anchorage loss and accepted heavy traction forces.

Retraction of anterior teeth can be achieved either by en-masse retraction, moving all the six anterior teeth together in a single step or by two-step retraction, separately retract canines in first step followed by retracting the four anteriors in the second step.

This Randomized Control Trial will be conducted to compare the effects of en-masse retraction to two- steps retraction on sagittal, vertical and dental dimensions using mini-implant as anchorage. 80 patients will be included in this study after meeting the eligibility criteria. Each group will contain 40 patients.

The patients will be divided in two groups i.e. two-step retraction group (control group) and en-masse group (experimental group), through software generated randomization table.

Two-step retraction group (control group) In this group, immediately after placement of mini-implant and extractions of upper first premolars, heavy ligation will be done from mini-implant to maxillary second premolar and first molar. Canine will be retracted by sliding mechanics and the four anterior teeth will be retracted by loop mechanics. Loops will be activated every three weeks by 1 mm.

Retraction will be stopped when canines establish class I relationship and a good incisor relationship will be obtained in both the groups

En-masse retraction group(experimental group) After placement of mini-implants and extraction of maxillary first premolar, rectangular stainless steel arch wire with anterior 8mm height crimpable hooks distal to the lateral incisors will be inserted and force will be applied using elastic chains attached between the mini-implant and the hooks for conducting en-masse retraction. Elastic chains will replace after every three weeks.

Pretreatment lateral cepalogram will be taken at time of enrolment (T1) and post-treatment lateral cephalogram taken after 12 months of orthodontic treatment (T2). All cephalometric radiograph will be traced on acetate tracing sheets 0.5 μm in thickness using a sharp 4H pencil on a view box using transilluminated light in a dark room.

The analysis will be done on pretreatment cephalogram (T1) and post treatment lateral cephalogram (T2) and then their measurements will be compared to find out changes in the sagittal, vertical and dental dimensions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both male and female patients with age of 18- 25 years. 2. Cases treated with upper first premolars extractions. 3. Cases having class II molar relation which is mesiobuccal cusp of maxillary first permanent molar occludes anterior to the buccal groove of mandibular first molar on both sides as assessed clinically.

  4. Overjet > 5mm and < 12mm as assessed clinically. 5. Cases with no remaining growth as assessed by cervical vertebrae maturation stages (cvm) ≥4 on lateral cephalometric radiograph .

  6. Cases with no congenitally missing teeth (excluding third molars).

Exclusion Criteria:

* 1. Long term use of systemic corticosteroids, calcium channel blockers & anti-inflammatory drugs.

  2. Cases with syndromes like cleft lip and palate as assessed clinically. 3. Cases in which active growth is still taking place as assessed by cervical vertebrae maturation stages (cvm) ≤ 3 on lateral cephalometric radiograph.

  4. Radiographic evidence of bone loss. 5. Periodontal disease as assessed clinically.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
To compare sagittal, vertical and dental dimensions following en-masse retraction with two-step retraction using mini-implants as anchorage. | Pretreatment lateral cepalogram will be taken at time of enrolment (T1) and post-treatment lateral cephalogram taken after 12 months of orthodontic treatment (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Anam Sattar, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
sagittal, vertical and dental dimensions following en-masse retraction with two-step retraction will be compared using mini-implants as anchorage
Supporting Information: Study Protocol, SAP, CSR
Time Frame: at the completion of study